CLINICAL TRIAL: NCT04147767
Title: Randomised Control Cross-over Trial to Test How Dietary Plant Sterols Modify Tumour Promoting Capabilities of Non-tumour Host Cells in Volunteers With Elevated LDL-C
Brief Title: Plant Sterol INtervention for Cancer Prevention (PINC)
Acronym: PINC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, James Thorne, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: RD19/123502
Record Dates: First submitted 2019-10-21; First posted 2019-11-01 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Hypercholesterolemia; Breast Cancer; Obesity
Keywords: oxysterol; breast cancer; phytosterols; cholesterol metabolism
MeSH Terms: conditions — Hypercholesterolemia; Breast Neoplasms; Obesity

STUDY DESIGN:
Intervention Model Description: Enrolled participants will undergo 1:1 simple randomisation by the CI, to either Experimental arm or placebo arm.. Evaluations after intervention will be made at the end of the first 8 weeks of intervention (Day 56; 8th week) and at the end of the second 8 weeks intervention (Day 140; 20th week). Since a wash out period between the two food products consumption is provided, another evaluation after wash out period (Day 84; 12th week) will be performed. The wash out period consist in a 4 weeks food products free period, where will be ask to participants to maintain their usual dietary and life style habits excluding the consumption of any yoghurt drinks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All trial investigators will be blinded to the intervention, except for the CI. The CI will keep a record of interventions administrated. All trial participants and outcome assessors will be blinded to the intervention. Each food product has the same flavour and taste, as well as the same packaging to ensure blinding in maintained throughout study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phytosterols Arm (Experimental): The investigational food product "Cholesterol Reducing Strawberry Yogurt Drink (Tesco)" is a strawberry yogurt drink with added plant sterols. A 100g bottle (one serving) of cholesterol lowering strawberry yogurt drink contains 2g of free plant sterols. The magnitude of the effect given by this enriched food product, providing a daily intake of 1,5-2,4 g plant sterols/stanols, refers to the lowering/reducing blood cholesterol effects in the range "7 % to 10 %" within 2 to 3 weeks of treatment, as specified by Commission Regulation (EU) 384/2010 of 05/05/2010.
  The dietary intervention will consist in 8 weeks consumption of PSS enriched Yogurt Drink, which provide a daily PSS intake of 3.4g/100g bottle plant sterols ester equivalent to 2g/100g bottle of free plant sterols.
  Interventions: Dietary Supplement: Cholesterol Reducing Strawberry Yogurt Drink (Tesco Ltd)
- Placebo Arm (Placebo Comparator): The investigational food product "Low Fat Strawberry Yogurt Drinks (Morrisons)" is a strawberry flavoured yogurt drink with sweetener and sugar, vitamin C, B6 and D, British milk.
  Placebo intervention consists in 8 weeks consumption of PSS non-enriched Yogurt Drinks. The placebo intervention is needed for the study design chosen (randomized double-blind placebo-controlled cross-over clinical trial). Placebo will be used in order to determine the efficacy of PSS intervention, comparing the effects of the two compounds (PSS and placebo) in the same experimental conditions and then avoiding bias.
  Interventions: Dietary Supplement: Low Fat Strawberry Yogurt Drinks (Morrisons Ltd)

INTERVENTIONS:
Dietary Supplement: Cholesterol Reducing Strawberry Yogurt Drink (Tesco Ltd) — Ingredients: Skimmed Milk, Strawberry Juice from Concentrate (5%), Plant Sterols Ester (3.4%)***, Sugar, Maize Starch, Flavourings, Colour (Anthocyanins), Starter Culture including Bifidobacterium (Milk), Thickener (Carob Gum), Sweetener (Sucralose), Milk Proteins.
  *** Equivalent to 2% Free Plant Sterols
  Arms: Phytosterols Arm
Dietary Supplement: Low Fat Strawberry Yogurt Drinks (Morrisons Ltd) — Ingredients: Yogurt (Milk), Water, Sugar, Strawberry Purée (1%), Modified Maize Starch, Carrot Concentrate, Flavouring, Acidity Regulator (Citric Acid), Vitamin C, Colour (Paprika Extract), Sweetener (Sucralose), Vitamin D, Vitamin B6.
  Arms: Placebo Arm

SUMMARY:
Several types of human cells convert cholesterol into other molecules, including oxysterols. Oxysterols can promote breast cancer growth and help tumours to spread. Some breast cancer types recruit other cells (host cells) able to produce oxysterols within the local cancer environment.

How these other cells help breast tumours metastasize or resist chemotherapy is not well understood, but epidemiological and clinical studies suggest elevated LDL-C is associated with worse survival, poorer response to therapy and an increased propensity for disease relapse in breast cancer patients. In this trial the investigators will test how an LDL-C lowering dietary intervention (using commercially available phytosterol added food products), alters the ability of non-cancer cells (adipocytes, fibroblasts and macrophages) collected from high LDL-C volunteers to change chemotherapy response and metastatic process in breast cancer cells.

In this trial, volunteers with high LDL-C levels will be recruited by the University of Leeds, and divided randomly into two arms that cross over. The experimental period (yogurt drink enriched with phytosterols) and placebo period (non-enriched yogurt drink) will each last for 8 weeks, alternated with a 4 weeks of wash-out period. Samples will be collected 4 times (week-0, week-8, week-12, week-20) during the study and will include blood, white blood cells (macrophages), and fat tissue cells. Measurements will include oxysterol, LDL-C and phytosterol concentrations (volunteers' serum/plasma, media from the host cells/breast cancer experimental culture) and how the host cells alter the behaviour of cancer cells in the laboratory.

DETAILED DESCRIPTION:
Delivery of cholesterol to extra-hepatic tissues by LDL has a profound impact on different host cell types, many of which themselves have been implicated in BCa metastasis and chemoresistance.

Despite accumulating data, it is still unknown how host-cells help breast tumours metastasise or evade chemotherapy. The molecular link between cholesterol and metastasis may involve the enzymatic hydroxylation (an intermediate step in bile acid synthesis) of cholesterol. The synthesis and secretion of oxysterols into the tumour microenvironment and this is exacerbated in individuals with elevated LDL-cholesterol. This process, occurring largely in macrophages, adipocytes and fibroblasts, leads to biosynthesis and cellular export of oxysterols , which drive DNA mutations through oxidative stress, confer resistance to chemotherapy, enhance BCa growth and metastasis, and are elevated in serum of BCa patients at metastatic relapse. Our pilot data show non-cancer host-cells activate oxysterols signalling and drug resistance protein expression and confer chemotherapy resistance in adjacent cancer cells.

The investigators therefore propose to test the hypothesis that the reason epidemiological and clinical studies find elevated LDL-C and its co-morbidities associate with worse survival in BCa patients, is because the host-cells of these patients have enhanced cholesterol metabolic flux leading to increased oxysterols production and improved tolerance of chemotherapy and promotion of cancer metastatic pathways.

This trial is a multicentre cross-over double blind clinical trial in which volunteers with LDL-C ≥160mg/dL (4.1 mmol/L), recruited at the University of Leeds and/or identified through Horizon 2020 project PATHWAY-27, will be randomised into two arms of intervention, Group A (experimental arm) will be given an yoghurt drink enriched with PSS and Group B (placebo comparator) will be given yoghurt drink non-enriched with PSS. Each dietary intervention will last for 8 weeks, alternated with a 4 weeks of wash out period. This trial wants to highlight the superiority of the PSS (yoghurt drink enriched) to placebo (yoghurt drink non-enriched) intervention on the improvement of the serum/plasma and host cells (adipocytes and macrophages) LDL-C, oxysterols , PSS levels in high LDL-C levels volunteers and in respective conditioned media from the host cells/BCa cell lines co-culture, and superiority of the PSS to placebo intervention on the improvement of the cholesterol panel levels involved in BCa tolerance of chemotherapy and metastatic progression, according also to the molecular and genetical pathways.

Because of the unknown effect of PSS on the oxysterols metabolism and of its consequent chemotherapy and anti-metastatic proprieties, the trial will be divided in two phases (I and II):

I. In this pilot phase the investigators will explore the effects of PSS intervention in 10 volunteers, evaluate feasibility of study protocol (participant recruitment and retention), and changes in mean and SD in oxysterols /PSS concentrations making changes to dose and power calculations if necessary. If the intervention causes any noteworthy effect in oxysterols serum/blood levels and/or on host cell co-culture with BCa cells the study will continue to Phase II:

II. In this phase a further 40 volunteers will be enrolled in the study satisfying our power calculation prediction to observe an effect.

This randomized cross-over double blind clinical trial will be run mainly at the School of Food Science and Nutrition, of the University of Leeds (FS&N). Each site will have a nominated principle investigator. This will be in collaboration with the NHS - Leeds Teaching Hospitals Trust (LTHT), the Leeds Institute of Biomedical & Clinical Sciences of the Faculty of Medicine and Health of the University of Leeds (LIBACS) and the Department of Chemistry of the University of Oslo (DC).

At each step point (Day 56, day 84 and day 140), the following trial assessments and procedures will be taken:

* Weight measurement;
* Participants diary card checking;
* Adverse effects and safety;
* Blood Pressure;
* Food intervention compliance checking by asking participants to return yoghurt packages back to trial team and relative recordings;
* 24h dietary recall questionnaire interview;
* LDL-C, HDL-C, Total Cholesterol, Triglycerides, non-HDL-C blood concentration and HDL-C/LDL-C ratio measurement;
* Serum/plasma OHCs concentration measurement;
* Serum/plasma PSS concentration measurement;
* Medium LDL-C concentration measurement after host cells co-culture with breast cancer cell lines;
* Medium OHCs concentration measurement after host cells co-culture with breast cancer cell lines;
* Medium PSS concentration measurement after host cells co-culture with breast cancer cell lines;
* Adipocytes, macrophages and breast cancer cell lines cell lines OHCs content measurement;
* Migratory and chemoresistance properties of the breast cancer cell lines cell lines after host cells co-culture.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects capable of giving informed consent;
2. Non-pregnant, non-nursing female;
3. Age between 18-65 years old;
4. LDL-C ≥130mg/dL (3.4mmol/L) or TC/HDL ratio >4;
5. BMI ≥25 (kg/m2)

Exclusion Criteria:

1. Subjects who are under treatment with lipophilic statins;
2. Subjects under any other supplementation that improve cholesterol levels (i.e. monacolin, other PSS enriched products);
3. Subjects under any weight loss or lipid lowering dietary plan;
4. Present or past chronic diseases: CVDs, cancer, know positive hepatitis B virus surface antigen (HBsAg), hepatitis C (HCV) antibody or HIV, cirrhosis, gastrointestinal disorders (i.e. irritable bowel syndrome, Crohn's disease, celiac disease, bowel control problems), kidney diseases, autoimmune diseases, endocrine disorders, metabolic diseases (i.e. diabetes type I and type II, familiar hypercholesterolemia), neurological diseases;
5. Diagnosed eating disorders according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5);
6. Past or planned within the trial period bariatric surgery;
7. Past or planned within the trial period gastrointestinal resections;
8. Corticosteroid and chronic inflammatory therapy;
9. Consumption within the preceding 8 weeks of other compounds capable of influencing cholesterol metabolism (bile acid-binding resins, ezetimibe, psyllium, fish oil supplements, soya lecithin, phytoestrogens and other PSS-fortified foods);
10. Females pregnant or females who are planning pregnancy;
11. Females breastfeeding;
12. Phytosterolemia diseases;
13. Participants with allergies to any of the substances presents in the yoghurt drink chosen for the trial: citric acid, anhydrous, sodium chloride, disodium edetate dehydrate, polysorbate 80, sodium hydroxide, Hypersensitivity to E. Coli derived proteins, nuts, peanuts, egg and soy proteins. Participants with a latex allergy are also not eligible as the inner needle cover of the pre-filled syringe contains dry natural rubber (a derivative of latex);
14. Participants with allergies to lidocaine;
15. Participation in other dietary or clinical trials.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To change circulating oxysterols levels after phytosterols intervention. | Serum/plasma oxysterols concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  The changes of oxysterols content in serum/plasma after 8 weeks of phytosterols intervention compared to placebo. After the dietary intervention, we expect to observe a change of -20% in circulating 27-hydroxycholesterol content (marker of oxysterols systemic levels).
  Concentration of oxysterols using LC-MS/MS measurement of plasma in 50 subjects after placebo and after intervention.

SECONDARY OUTCOMES:
Change intra-cellular adipocyte and macrophages oxysterols concentrations | Serum/plasma/medium oxysterols concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Concentration of oxysterols using LC-MS/MS measurement of host cells in 50 subjects after placebo and after intervention.
  Effect of phytosterols enriched foods consumption compared to placebo intervention on migratory and chemoresistance properties of breast cancer cell lines (MDA.MB.231, MDA.MB.468, MCF7 and T47D) when in co-culture with the host-cells collected in each step of the trial.
Study of adipocytes and macrophages interaction with breast cancer cell lines | Protein expression will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Effect of phytosterols enriched foods consumption compared to placebo intervention on migratory and chemoresistance properties of breast cancer cell lines (MDA.MB.231, MDA.MB.468, MCF7 and T47D) when in co-culture with the host-cells collected in each step of the trial.
  Changes in proteins expression of oxysterols target genes.
Study of adipocytes and macrophages interaction with breast cancer cell lines | Gene expression will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Effect of phytosterols enriched foods consumption compared to placebo intervention on migratory and chemoresistance properties of breast cancer cell lines (MDA.MB.231, MDA.MB.468, MCF7 and T47D) when in co-culture with the host-cells collected in each step of the trial.
  Changes in gene expression of oxysterols target genes.
Study the effect of phytosterols on LDL-C | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Study of the effect of phytosterols on LDL-C concentration in 50 subjects after placebo and after intervention using Alere Afinion™.
Study the effect of phytosterols on HDL-C | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Study of the effect of phytosterols on HDL-C concentration in 50 subjects after placebo and after intervention using Alere Afinion™.
Study the effect of phytosterols on Total Cholesterol | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Study of the effect of phytosterols on Total Cholesterol concentration in 50 subjects after placebo and after intervention using Alere Afinion™.
Study the effect of phytosterols on Triglycerides | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Study of the effect of phytosterols on Triglycerides concentration in 50 subjects after placebo and after intervention using Alere Afinion™.
Study the effect of phytosterols on non-HDL-C | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Study of the effect of phytosterols on non-HDL-C concentration in 50 subjects after placebo and after intervention using Alere Afinion™.
Quantify phytosterols in blood samples from volunteers. | Serum/plasma phytosterols and lipid concentrations will be measured during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Phytosterols panel serum/plasma levels after phytosterols enriched food or placebo intervention during all the steps of the trial.

OTHER OUTCOMES:
Study RNA sequences changes in the oxysterols/LDL-C pathway and secondary breast cancer before and after phytosterols intervention . | RNA will be studied during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  RNA sequence will be measured with RNA-seq techniques before and after phytosterols intervention to identify the molecular effectors of the paracrine regulatory systems in the oxysterols, LDL-C and secondary BCa pattern.
Study changes in the interactions between proteins and DNA in the oxysterols/LDL-C pathway and secondary breast cancer before and after phytosterols intervention . | interactions between proteins and DNA will be studied during all the steps of the trial (baseline, 8th week, 12nd week, 20th week)
  Changes in interactions between proteins and DNA and using Chip/seq will be measured before and after phytosterols intervention to identify the molecular effectors of the paracrine regulatory systems in the oxysterols, LDL-C and secondary BCa pattern.

CONTACTS AND LOCATIONS:
Overall Officials: James L Thorne, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in scientific journals, which will depend on the outcome of data analysis. Anonymized research data will be deposited with the University of Leeds data repository.